CLINICAL TRIAL: NCT00373685
Title: Gastrointestinal (GI) Randomized Event And Safety Open-Label NSAID Study (GI-Reasons): A Randomized, Open-Label, Blinded-Endpoint, Parallel-Group Trial Of GI Safety Of Celecoxib Compared With Non-Selective Nonsteroidal Antiinflammatory Drugs (NSAIDS) In Osteoarthritis Patients
Brief Title: GI-Reasons- A Trial Of GI Safety Of Celecoxib Compared With Non-Selective Nonsteroidal Antiinflammatory Drugs (NSAIDS)
Acronym: GI-REASONS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3191331
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
Keywords: GI events in patients with moderate GI risk treated with NSAIDS
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Experimental): dosing as per USPI label
  Interventions: Drug: Celecoxib
- NSAIDs (Active Comparator)
  Interventions: Drug: Any commercially available NSAID with the indication for osteoarthritis

INTERVENTIONS:
Drug: Celecoxib — open-label
  Arms: Celecoxib
Drug: Any commercially available NSAID with the indication for osteoarthritis — dosing as per USPI label related to the chosen commercially marketed NSAID
  Arms: NSAIDs

SUMMARY:
This study investigates if Celebrex has a lower incident of Gastrointestinal Events than other NSAIDS in subjects with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of at least 55 years of age with a clinical diagnosis of OA who are expected to require daily prescription anti-inflammatory analgesic therapy for arthritis symptom management and for whom either celecoxib or a nsNSAID is an appropriate treatment option.

Exclusion Criteria:

* GI ulcer hemorrhage or active GD ulceration less than 90 days prior to screening visit.
* Patients with a history of myocardial infarction, unstable angina, ischemic or hemorrhagic stroke, transient ischemic attack, previous revascularization procedure to coronary, carotid, cerebral, renal, aortic or peripheral arterial vasculature.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8067 (Actual)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (628):
- United States (606):
  - Pfizer Investigational Site, Abbeville, Alabama
  - Pfizer Investigational Site, Alexander City, Alabama
  - Pfizer Investigational Site, Bay Minette, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Cullman, Alabama
  - Pfizer Investigational Site, Dothan, Alabama
  - Pfizer Investigational Site, Geneva, Alabama
  - Pfizer Investigational Site, Gulf Shores, Alabama
  - Pfizer Investigational Site, Guntersville, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Jacksonville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Muscle Shoals, Alabama
  - Pfizer Investigational Site, Ozark, Alabama
  - Pfizer Investigational Site, Pell City, Alabama
  - Pfizer Investigational Site, Tallassee, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Green Valley, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Sierra Vista, Arizona
  - Pfizer Investigational Site, Sun Lakes, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Paragould, Arkansas
  - Pfizer Investigational Site, Pine Bluff, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Bellflower, California
  - Pfizer Investigational Site, Bermuda Dunes, California
  - Pfizer Investigational Site, Buena Park, California
  - Pfizer Investigational Site, Carson, California
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Cudahy, California
  - Pfizer Investigational Site, El Cajon, California
  - Pfizer Investigational Site, El Segundo, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Fortuna, California
  - Pfizer Investigational Site, Fremont, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Harbor City, California
  - Pfizer Investigational Site, Hemet, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Huntington Park, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, La Palma, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Los Banos, California
  - Pfizer Investigational Site, Los Gatos, California
  - Pfizer Investigational Site, Marina del Rey, California
  - Pfizer Investigational Site, Merced, California
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Montebello, California
  - Pfizer Investigational Site, Monterey Park, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Rancho Cucamonga, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, Reseda, California
  - Pfizer Investigational Site, Rialto, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Rowland Heights, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, San Leandro, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Santa Maria, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Tulare, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Van Nuys, California
  - Pfizer Investigational Site, Victorville, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Westminster, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Wildomar, California
  - Pfizer Investigational Site, Wilmington, California
  - Pfizer Investigational Site, Woodland Hills, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Fort Collins, Colorado
  - Pfizer Investigational Site, Golden, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Northglenn, Colorado
  - Pfizer Investigational Site, Pueblo, Colorado
  - Pfizer Investigational Site, Avon, Connecticut
  - Pfizer Investigational Site, Brewster, Connecticut
  - Pfizer Investigational Site, Brookfield, Connecticut
  - Pfizer Investigational Site, Cos Cob, Connecticut
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Milford, Connecticut
  - Pfizer Investigational Site, Ridgefield, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Smyrna, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Apopka, Florida
  - Pfizer Investigational Site, Beverly Hills, Florida
  - Pfizer Investigational Site, Boynton Beach, Florida
  - Pfizer Investigational Site, Chipley, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Clermont, Florida
  - Pfizer Investigational Site, Cocoa, Florida
  - Pfizer Investigational Site, Cocoa Beach, Florida
  - Pfizer Investigational Site, Coral Springs, Florida
  - Pfizer Investigational Site, Crystal River, Florida
  - Pfizer Investigational Site, Cutler Bay, Florida
  - Pfizer Investigational Site, Davie, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Dunnellon, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Green Cove Springs, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Hialeah, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Key Biscayne, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Niceville, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Oviedo, Florida
  - Pfizer Investigational Site, Palm Bay, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Panama City, Florida
  - Pfizer Investigational Site, Parkland, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Pinecrest, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Port Orange, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, Saint Cloud, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Sebastian, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Wellington, Florida
  - Pfizer Investigational Site, Athens, Georgia
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Bainbridge, Georgia
  - Pfizer Investigational Site, Cairo, Georgia
  - Pfizer Investigational Site, Calhoun, Georgia
  - Pfizer Investigational Site, Cartersville, Georgia
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Covington, Georgia
  - Pfizer Investigational Site, Cumming, Georgia
  - Pfizer Investigational Site, Dawsonville, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Dunwoody, Georgia
  - Pfizer Investigational Site, Gainesville, Georgia
  - Pfizer Investigational Site, Hampton, Georgia
  - Pfizer Investigational Site, Hinesville, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Roswell, Georgia
  - Pfizer Investigational Site, Sandersville, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Snellville, Georgia
  - Pfizer Investigational Site, Stockbridge, Georgia
  - Pfizer Investigational Site, Watkinsville, Georgia
  - Pfizer Investigational Site, Waycross, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, ‘Aiea, Hawaii
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Danville, Illinois
  - Pfizer Investigational Site, DeKalb, Illinois
  - Pfizer Investigational Site, Elgin, Illinois
  - Pfizer Investigational Site, Evergreen Park, Illinois
  - Pfizer Investigational Site, Fairview Heights, Illinois
  - Pfizer Investigational Site, Flossmoor, Illinois
  - Pfizer Investigational Site, Greenville, Illinois
  - Pfizer Investigational Site, Hanna City, Illinois
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Moweaqua, Illinois
  - Pfizer Investigational Site, O'Fallon, Illinois
  - Pfizer Investigational Site, Pekin, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Quincy, Illinois
  - Pfizer Investigational Site, Watseka, Illinois
  - Pfizer Investigational Site, Brownsburg, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Hobart, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, La Porte, Indiana
  - Pfizer Investigational Site, Mishawaka, Indiana
  - Pfizer Investigational Site, New Haven, Indiana
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Wabash, Indiana
  - Pfizer Investigational Site, Ames, Iowa
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Fort Dodge, Iowa
  - Pfizer Investigational Site, Waterloo, Iowa
  - Pfizer Investigational Site, West Burlington, Iowa
  - Pfizer Investigational Site, Arkansas City, Kansas
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Mission, Kansas
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Wellington, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Bowling Green, Kentucky
  - Pfizer Investigational Site, Draffenville, Kentucky
  - Pfizer Investigational Site, Hartford, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Paducah, Kentucky
  - Pfizer Investigational Site, Richmond, Kentucky
  - Pfizer Investigational Site, Alexandria, Louisiana
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Jena, Louisiana
  - Pfizer Investigational Site, Jonesboro, Louisiana
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Monroe, Louisiana
  - Pfizer Investigational Site, Natchitoches, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bel Air, Maryland
  - Pfizer Investigational Site, Bladensburg, Maryland
  - Pfizer Investigational Site, College Park, Maryland
  - Pfizer Investigational Site, Elkton, Maryland
  - Pfizer Investigational Site, Ellicott City, Maryland
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Mount Airy, Maryland
  - Pfizer Investigational Site, Prince Frederick, Maryland
  - Pfizer Investigational Site, Riverdale, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Silver Spring, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Attleboro, Massachusetts
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, North Andover, Massachusetts
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Taunton, Massachusetts
  - Pfizer Investigational Site, Berkley, Michigan
  - Pfizer Investigational Site, Brighton, Michigan
  - Pfizer Investigational Site, Cadillac, Michigan
  - Pfizer Investigational Site, Chelsea, Michigan
  - Pfizer Investigational Site, Clarkston, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Fair Haven, Michigan
  - Pfizer Investigational Site, Fenton, Michigan
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Grand Ledge, Michigan
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Interlochen, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Parchment, Michigan
  - Pfizer Investigational Site, Pigeon, Michigan
  - Pfizer Investigational Site, Saginaw, Michigan
  - Pfizer Investigational Site, Saint Clair Shores, Michigan
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Southgate, Michigan
  - Pfizer Investigational Site, Sterling Heights, Michigan
  - Pfizer Investigational Site, Sturgis, Michigan
  - Pfizer Investigational Site, Traverse City, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, West Branch, Michigan
  - Pfizer Investigational Site, Ypsilanti, Michigan
  - Pfizer Investigational Site, Belzoni, Mississippi
  - Pfizer Investigational Site, Hattiesburg, Mississippi
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Magee, Mississippi
  - Pfizer Investigational Site, Picayune, Mississippi
  - Pfizer Investigational Site, Port Gibson, Mississippi
  - Pfizer Investigational Site, Prentiss, Mississippi
  - Pfizer Investigational Site, Sumrall, Mississippi
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Florissant, Missouri
  - Pfizer Investigational Site, Jackson, Missouri
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Missoula, Montana
  - Pfizer Investigational Site, Alliance, Nebraska
  - Pfizer Investigational Site, Beatrice, Nebraska
  - Pfizer Investigational Site, Broken Bow, Nebraska
  - Pfizer Investigational Site, Fremont, Nebraska
  - Pfizer Investigational Site, Grand Island, Nebraska
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, McCook, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Incline Village, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Belvidere, New Jersey
  - Pfizer Investigational Site, Berlin, New Jersey
  - Pfizer Investigational Site, Blackwood, New Jersey
  - Pfizer Investigational Site, Bridgeport, New Jersey
  - Pfizer Investigational Site, Bridgeton, New Jersey
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Egg Harbor, New Jersey
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Flanders, New Jersey
  - Pfizer Investigational Site, Freehold, New Jersey
  - Pfizer Investigational Site, Glendora, New Jersey
  - Pfizer Investigational Site, Holmdel, New Jersey
  - Pfizer Investigational Site, Lincoln Park, New Jersey
  - Pfizer Investigational Site, Linden, New Jersey
  - Pfizer Investigational Site, Midland Park, New Jersey
  - Pfizer Investigational Site, North Arlington, New Jersey
  - Pfizer Investigational Site, Passaic, New Jersey
  - Pfizer Investigational Site, South Bound Brook, New Jersey
  - Pfizer Investigational Site, Voorhees Township, New Jersey
  - Pfizer Investigational Site, Whitehouse Station, New Jersey
  - Pfizer Investigational Site, Wildwood Crest, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Los Alamos, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, East Syracuse, New York
  - Pfizer Investigational Site, Elmhurst, New York
  - Pfizer Investigational Site, Far Rockaway, New York
  - Pfizer Investigational Site, Fayetteville, New York
  - Pfizer Investigational Site, Flushing, New York
  - Pfizer Investigational Site, Forest Hills, New York
  - Pfizer Investigational Site, Lake Success, New York
  - Pfizer Investigational Site, Lewiston, New York
  - Pfizer Investigational Site, Liverpool, New York
  - Pfizer Investigational Site, New Hartford, New York
  - Pfizer Investigational Site, New Windsor, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Plainview, New York
  - Pfizer Investigational Site, Rye Brook, New York
  - Pfizer Investigational Site, Salamanca, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Tonawanda, New York
  - Pfizer Investigational Site, Wantagh, New York
  - Pfizer Investigational Site, Warsaw, New York
  - Pfizer Investigational Site, West Babylon, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Asheboro, North Carolina
  - Pfizer Investigational Site, Boone, North Carolina
  - Pfizer Investigational Site, Bunn, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Elizabeth City, North Carolina
  - Pfizer Investigational Site, Gastonia, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Jacksonville, North Carolina
  - Pfizer Investigational Site, Kinston, North Carolina
  - Pfizer Investigational Site, Lenoir, North Carolina
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, New Bern, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Shelby, North Carolina
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Tabor City, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Boardman, Ohio
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Carlisle, Ohio
  - Pfizer Investigational Site, Centerville, Ohio
  - Pfizer Investigational Site, Chardon, Ohio
  - Pfizer Investigational Site, Chesterland, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Cortland, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Delaware, Ohio
  - Pfizer Investigational Site, Fairborn, Ohio
  - Pfizer Investigational Site, Franklin, Ohio
  - Pfizer Investigational Site, Genoa, Ohio
  - Pfizer Investigational Site, Lyndhurst, Ohio
  - Pfizer Investigational Site, Marietta, Ohio
  - Pfizer Investigational Site, Marion, Ohio
  - Pfizer Investigational Site, Mason, Ohio
  - Pfizer Investigational Site, McConnelsville, Ohio
  - Pfizer Investigational Site, Middleburg Heights, Ohio
  - Pfizer Investigational Site, Middletown, Ohio
  - Pfizer Investigational Site, New Lexington, Ohio
  - Pfizer Investigational Site, Orrville, Ohio
  - Pfizer Investigational Site, Shaker Heights, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Trenton, Ohio
  - Pfizer Investigational Site, Wadsworth, Ohio
  - Pfizer Investigational Site, Warren, Ohio
  - Pfizer Investigational Site, Westlake, Ohio
  - Pfizer Investigational Site, Willoughby Hills, Ohio
  - Pfizer Investigational Site, Wooster, Ohio
  - Pfizer Investigational Site, Zanesville, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Edmond, Oklahoma
  - Pfizer Investigational Site, Moore, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Stillwater, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Yukon, Oklahoma
  - Pfizer Investigational Site, Grants Pass, Oregon
  - Pfizer Investigational Site, Hermiston, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Aston Mills, Pennsylvania
  - Pfizer Investigational Site, Audubon, Pennsylvania
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Bristol, Pennsylvania
  - Pfizer Investigational Site, Broomall, Pennsylvania
  - Pfizer Investigational Site, Butler, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Carnegie, Pennsylvania
  - Pfizer Investigational Site, Chester, Pennsylvania
  - Pfizer Investigational Site, Chicora, Pennsylvania
  - Pfizer Investigational Site, Cresson, Pennsylvania
  - Pfizer Investigational Site, Dallastown, Pennsylvania
  - Pfizer Investigational Site, Dauphin, Pennsylvania
  - Pfizer Investigational Site, Downingtown, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Erie, Pennsylvania
  - Pfizer Investigational Site, Fleetwood, Pennsylvania
  - Pfizer Investigational Site, Flourtown, Pennsylvania
  - Pfizer Investigational Site, Fogelsville, Pennsylvania
  - Pfizer Investigational Site, Greensburg, Pennsylvania
  - Pfizer Investigational Site, Harrisburg, Pennsylvania
  - Pfizer Investigational Site, Hatboro, Pennsylvania
  - Pfizer Investigational Site, Hatfield, Pennsylvania
  - Pfizer Investigational Site, Jeannette, Pennsylvania
  - Pfizer Investigational Site, Jefferson Hills, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, King of Prussia, Pennsylvania
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Millvale, Pennsylvania
  - Pfizer Investigational Site, Morrisville, Pennsylvania
  - Pfizer Investigational Site, Northern Cambria, Pennsylvania
  - Pfizer Investigational Site, Penndel, Pennsylvania
  - Pfizer Investigational Site, Pennsburg, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Phoenixville, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Port Carbon, Pennsylvania
  - Pfizer Investigational Site, Pottstown, Pennsylvania
  - Pfizer Investigational Site, Reading, Pennsylvania
  - Pfizer Investigational Site, Scranton, Pennsylvania
  - Pfizer Investigational Site, Thorndale, Pennsylvania
  - Pfizer Investigational Site, Tipton, Pennsylvania
  - Pfizer Investigational Site, Uniontown, Pennsylvania
  - Pfizer Investigational Site, Upper Saint Clair, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Zionsville, Pennsylvania
  - Pfizer Investigational Site, Cranston, Rhode Island
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Bluffton, South Carolina
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Clemson, South Carolina
  - Pfizer Investigational Site, Clinton, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Gaffney, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Landrum, South Carolina
  - Pfizer Investigational Site, Marion, South Carolina
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Newberry, South Carolina
  - Pfizer Investigational Site, North Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Peak, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Taylors, South Carolina
  - Pfizer Investigational Site, Union, South Carolina
  - Pfizer Investigational Site, Bolivar, Tennessee
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Clarksville, Tennessee
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Hendersonville, Tennessee
  - Pfizer Investigational Site, Humboldt, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Maynardville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Morristown, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Springfield, Tennessee
  - Pfizer Investigational Site, Amarillo, Texas
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Azle, Texas
  - Pfizer Investigational Site, Carrollton, Texas
  - Pfizer Investigational Site, Colleyville, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Farmers Branch, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Frisco, Texas
  - Pfizer Investigational Site, Garland, Texas
  - Pfizer Investigational Site, Grand Prairie, Texas
  - Pfizer Investigational Site, Grapevine, Texas
  - Pfizer Investigational Site, Henderson, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Humble, Texas
  - Pfizer Investigational Site, Hurst, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Katy, Texas
  - Pfizer Investigational Site, Killeen, Texas
  - Pfizer Investigational Site, McKinney, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, Missouri City, Texas
  - Pfizer Investigational Site, Nederland, Texas
  - Pfizer Investigational Site, New Braunfels, Texas
  - Pfizer Investigational Site, North Richland Hills, Texas
  - Pfizer Investigational Site, Odessa, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Pleasanton, Texas
  - Pfizer Investigational Site, Poteet, Texas
  - Pfizer Investigational Site, Richardson, Texas
  - Pfizer Investigational Site, Richmond, Texas
  - Pfizer Investigational Site, Rockwall, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Seguin, Texas
  - Pfizer Investigational Site, Southlake, Texas
  - Pfizer Investigational Site, Spring, Texas
  - Pfizer Investigational Site, Stephenville, Texas
  - Pfizer Investigational Site, Sugar Land, Texas
  - Pfizer Investigational Site, Sulphur Springs, Texas
  - Pfizer Investigational Site, The Woodlands, Texas
  - Pfizer Investigational Site, Tomball, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Clinton, Utah
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, St. George, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Annandale, Virginia
  - Pfizer Investigational Site, Bluefield, Virginia
  - Pfizer Investigational Site, Chatham, Virginia
  - Pfizer Investigational Site, Chesapeake, Virginia
  - Pfizer Investigational Site, Danville, Virginia
  - Pfizer Investigational Site, Hampton, Virginia
  - Pfizer Investigational Site, Honaker, Virginia
  - Pfizer Investigational Site, Leesburg, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Portsmouth, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Vienna, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Pasco, Washington
  - Pfizer Investigational Site, Selah, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Walla Walla, Washington
  - Pfizer Investigational Site, Burnsville, West Virginia
  - Pfizer Investigational Site, Lewisburg, West Virginia
  - Pfizer Investigational Site, Ronceverte, West Virginia
- Puerto Rico (22):
  - Pfizer Investigational Site, Aguas Buenas, PR
  - Pfizer Investigational Site, Aguns Buenoas, PR
  - Pfizer Investigational Site, Aibonito, PR
  - Pfizer Investigational Site, Bayamón, PR
  - Pfizer Investigational Site, Caguas, PR
  - Pfizer Investigational Site, Carolina, PR
  - Pfizer Investigational Site, Cayey, PR
  - Pfizer Investigational Site, Cialis, PR
  - Pfizer Investigational Site, Cidra, PR
  - Pfizer Investigational Site, Hato Rey, PR
  - Pfizer Investigational Site, Juncas, PR
  - Pfizer Investigational Site, Juncos, PR
  - Pfizer Investigational Site, Las Piedras, PR
  - Pfizer Investigational Site, Levittown, PR
  - Pfizer Investigational Site, Manatí, PR
  - Pfizer Investigational Site, Rio Piedras, PR
  - Pfizer Investigational Site, San Juan, PR
  - Pfizer Investigational Site, Santa Isabel, PR
  - Pfizer Investigational Site, Santurce, PR
  - Pfizer Investigational Site, Trujillo Alto, PR
  - Pfizer Investigational Site, Loíza
  - Pfizer Investigational Site, Orocovis

REFERENCES:
- [Derived] Cryer B, Li C, Simon LS, Singh G, Stillman MJ, Berger MF. GI-REASONS: a novel 6-month, prospective, randomized, open-label, blinded endpoint (PROBE) trial. Am J Gastroenterol. 2013 Mar;108(3):392-400. doi: 10.1038/ajg.2012.467. Epub 2013 Feb 12. PMID 23399552
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191331&StudyName=GI-Reasons-%20A%20Trial%20Of%20GI%20Safety%20Of%20Celecoxib%20Compared%20With%20Non-Selective%20Nonsteroidal%20Antiinflammatory%20Drugs%20%28NSAIDS%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 8140 participants were randomized into the trial, however the final analysis was on 8067 participants because 35 participants were randomized twice and 1 participant was randomized 3 times, totaling 73.
Groups:
- Celecoxib: Celecoxib open-label per United States Package Insert (US PI) recommended dosing
- nsNSAIDs: Prescription non-selective nonsteroidal anti-inflammatory drug (nsNSAID) treatment (except for aspirin), per US PI recommended dosing
Period: Overall Study
Arm/Group | Celecoxib | nsNSAIDs
Started | 4035 | 4032
Treated | 3984 | 3955
Completed | 2596 | 2611
Not Completed | 1439 | 1421
Not completed — Death | 2 | 1
Not completed — Adverse Event | 278 | 253
Not completed — Insufficient clinical response | 169 | 119
Not completed — Did not meet entrance criteria | 167 | 184
Not completed — Lost to follow up | 83 | 103
Not completed — No longer willing to participate | 337 | 352
Not completed — Other | 149 | 146
Not completed — Protocol Violation | 191 | 182
Not completed — Final Status Unknown | 12 | 4
Not completed — Randomized, not treated | 51 | 77

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | nsNSAIDs | Total
Number analyzed (Participants) | 4035 | 4032 | 8067
Age, Customized [Number; unit: Participants]
  <55 years | 5 | 2 | 7
  55-59 years | 1339 | 1361 | 2700
  60-64 years | 1149 | 1127 | 2276
  65-69 years | 848 | 822 | 1670
  70-74 years | 504 | 517 | 1021
  >=75 years | 184 | 197 | 381
  Unspecified | 6 | 6 | 12
Sex/Gender, Customized [Number; unit: Participants]
  Male | 980 | 962 | 1942
  Female | 3049 | 3064 | 6113
  Unspecified | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Upper and/or Lower Gastrointestinal Events (CSULGIEs)
Description: CSULGIE defined as any of the following: gastroduodenal (GD) hemorrhage; gastric outlet obstruction; GD, small or large bowel perforation; small or large bowel hemorrhage; acute gastrointestinal (GI) hemorrhage of unknown origin; small bowel obstruction; clinically significant anemia/blood loss of defined GI origin or presumed occult GI origin.
Time Frame: Baseline through week 24 or Early Termination (ET)
Population: Intent-to-Treat (ITT) Population: randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 4035 | 4032
Percentage of participants | 1.3 | 2.4
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Test type: Superiority or Other; p = 0.0003, Life Table Extension of CMH Test — Life Table Extension of Cochran-Mantel-Haenszel (CMH) Test

2. Secondary Outcome: Percentage of Participants With Moderate to Severe Abdominal Symptoms
Description: Abdominal symptoms coded using the Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) 'Gastrointestinal Disorders' high level group term (HLGT) equal to "Gastrointestinal Signs and Symptoms"; where moderate indicated the gastrointestinal adverse event (GI AE) interfered to some extent with the participants' usual function and severe indicated the GI AE interfered significantly with participants' usual function.
Time Frame: Baseline through week 24 or ET
Population: ITT;
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 4035 | 4032
Percentage of participants | 2.3 | 3.4
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Test type: Superiority or Other; p = 0.0035, Life Table Extension of CMH Test

3. Secondary Outcome: Percentage of Participants Who Withdrew Due to GI Adverse Events (AEs)
Description: GI AEs defined using MedDRA SOC 'Gastrointestinal Disorders' but excluding HLGT's: Benign Neoplasms Gastrointestinal, Dental and Gingival Conditions, Oral Soft Tissue Conditions, Salivary Gland Conditions and Tongue Conditions
Time Frame: Baseline through week 24 or ET
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 4035 | 4032
Percentage of participants | 2.8 | 3.0
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Test type: Superiority or Other; p = 0.6140, Life Table Extension of CMH Test

4. Secondary Outcome: Hemoglobin (Hb) at Baseline
Time Frame: Baseline
Population: ITT; N= number of evaluable participants analyzed
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3604 | 3574
gram per deciliter (g/dL) | 13.6 (1.1) | 13.6 (1.2)

5. Secondary Outcome: Change From Baseline Hb at Week 24
Time Frame: Baseline and Week 24 or ET
Population: ITT; N=number of evaluable participants analyzed; Last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3604 | 3574
g/dL | -0.109 (0.012) | -0.241 (0.012)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value associated with Overall (LOCF)

6. Secondary Outcome: Hematocrit (Hct) at Baseline
Time Frame: Baseline
Population: ITT; N= number of evaluable participants analyzed
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3596 | 3568
Percent | 40.8 (3.4) | 40.9 (3.4)

7. Secondary Outcome: Change From Baseline Hct at Week 24
Time Frame: Baseline and Week 24 or ET
Population: ITT; N= number of evaluable participants analyzed; LOCF
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3596 | 3568
Percent | -0.330 (0.038) | -0.716 (0.039)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value associated with Overall (LOCF)

8. Secondary Outcome: Percentage of Participants With Clinically Significant Decrease in Hct and/or Hb From Baseline
Description: Clinically significant decrease in Hct (greater than or equal to 10 percent [≥10%]) and/or decrease in Hb (≥ 2 g/dL).
Time Frame: Baseline, Weeks 8, 16, 24 or ET
Population: ITT; N=number of evaluable participants analyzed; n=number of evaluable participants analyzed at the specific time point; LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3604 | 3574
Percentage of participants
  Week 8 (n= 3043, 3086) | 0.7 | 0.9
  Week 16 (n=2687, 2675) | 0.8 | 1.6
  Week 24 (n=3278, 3207) | 0.9 | 1.5
  Week 24 LOCF (n=3604, 3574) | 1.8 | 2.9
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Test type: Superiority or Other; p = 0.0023, Cochran-Mantel-Haenszel — P-value associated with Overall (LOCF)

9. Secondary Outcome: Percentage of Participants Satisfied With Efficacy of Current Pain Medication Overall
Description: Percentage of participants who reported Very Satisfied or Satisfied with current pain medication question on the Patient Treatment Satisfaction Scale (PTSS), scale ranged from Very Satisfied (1) to Very Dissatisfied (5).
Time Frame: Baseline, Weeks 8, 16, 24 or ET
Population: ITT; N=number of evaluable participants analyzed; n=number of evaluable participants analyzed at specific time point; LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3887 | 3904
Percentage of participants
  Baseline (n=3887, 3904) | 39.8 | 38.0
  Week 8 (n=3181, 3199) | 78.5 | 69.5
  Week 16 (n=2784, 2772) | 81.9 | 74.6
  Week 24 or ET (n=3383, 3361) | 74.6 | 70.8
  Week 24/LOCF (n=3672, 3651) | 74.5 | 70.3
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Baseline; Test type: Superiority or Other; p = 0.1008, Chi-squared
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Week 8; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Week 16; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Celecoxib vs nsNSAIDs; Week 24 or ET; Test type: Superiority or Other; p = 0.0005, Chi-squared
Statistical Analysis 5: Comparison: Celecoxib vs nsNSAIDs; Week 24/LOCF; Test type: Superiority or Other; p < 0.0001, Chi-squared

10. Secondary Outcome: Percentage of Participants Satisfied With Efficacy of Current Pain Medication - Time to Pain Relief
Description: Percentage of participants who reported Very Satisfied or Satisfied with efficacy of current pain medication questions on the PTSS Efficacy subscale for the time it took medication to work, scale ranged from Very Satisfied (1) to Very Dissatisfied (5). Possible range of scores 1 to 15.
Time Frame: Baseline, Weeks 8, 16, 24 or ET
Population: ITT; N=number of evaluable participants analyzed; n= number of evaluable participants analyzed at specific time point; LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3890 | 3905
Percentage of participants
  Baseline (n=3890, 3905) | 43.2 | 43.7
  Week 8 (n=3185, 3202) | 80.2 | 71.6
  Week 16 (n=2784,2777) | 83.2 | 77.7
  Week 24 or ET (n=3386,3362) | 76.2 | 73.8
  Week 24/LOCF (n=3672, 3653) | 76.0 | 73.3
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Baseline; Test type: Superiority or Other; p = 0.6562, Chi-squared
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Week 8; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Week 16; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Celecoxib vs nsNSAIDs; Week 24 or ET; Test type: Superiority or Other; p = 0.0245, Chi-squared
Statistical Analysis 5: Comparison: Celecoxib vs nsNSAIDs; Week 24/LOCF; Test type: Superiority or Other; p = 0.0074, Chi-squared

11. Secondary Outcome: Percentage of Participants Satisfied With Efficacy of Current Pain Medication - Amount of Pain Relief
Description: Percentage of participants who reported Very Satisfied or Satisfied with efficacy of current pain medication questions on the PTSS Efficacy subscale for the amount of pain relief medication provided, scale ranged from Very Satisfied (1) to Very Dissatisfied (5). Possible range of scores 1 to 15.
Time Frame: Baseline, Weeks 8, 16, 24 or ET
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3888 | 3905
Percentage of participants
  Baseline (n=3888, 3905) | 41.4 | 40.5
  Week 8 (n=3185, 3203) | 77.4 | 69.2
  Week 16 (n=2783, 2778) | 80.5 | 74.5
  Week 24 or ET (n=3385, 3362) | 74.0 | 71.3
  Week 24/LOCF (n=3671, 3653) | 74.0 | 70.8
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Baseline; Test type: Superiority or Other; p = 0.4074, Chi-squared
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Week 8; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Week 16; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Celecoxib vs nsNSAIDs; Week 24 or ET; Test type: Superiority or Other; p = 0.0127, Chi-squared
Statistical Analysis 5: Comparison: Celecoxib vs nsNSAIDs; Week 24/LOCF; Test type: Superiority or Other; p = 0.0019, Chi-squared

12. Secondary Outcome: Percentage of Participants Satisfied With Efficacy of Current Pain Medication - Duration of Pain Relief
Description: Percentage of participants who reported Very Satisfied or Satisfied with efficacy of current pain medication questions on the PTSS Efficacy, subscale for duration of pain relief provided by medication, scale ranged from Very Satisfied (1) to Very Dissatisfied (5). Possible range of scores 1 to 15.
Time Frame: Baseline, Weeks 8, 16, 24 or ET
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3886 | 3905
Percentage of participants
  Baseline (n=3886, 3905) | 37.8 | 36.6
  Week 8 (n=3182, 3202) | 75.4 | 66.8
  Week 16 (n=2780,2778) | 77.8 | 71.6
  Week 24 or ET (n=3383,3361) | 72.2 | 68.8
  Week 24/LOCF (n=3671, 3653) | 72.2 | 68.2
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Baseline; Test type: Superiority or Other; p = 0.2699, Chi-squared
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Week 8; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Week 16; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Celecoxib vs nsNSAIDs; Week 24 or ET; Test type: Superiority or Other; p = 0.0027, Chi-squared
Statistical Analysis 5: Comparison: Celecoxib vs nsNSAIDs; Week 24/LOCF; Test type: Superiority or Other; p = 0.0001, Chi-squared

13. Other Pre Specified Outcome: Percentage of Participants With Positive Blood Fecal Occult
Description: Positive blood fecal occult; blood in feces that is not visibly apparent
Time Frame: Week 24 or ET
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 4035 | 4032
Percentage of participants | 1.1 | 1.4

14. Other Pre Specified Outcome: Percentage of Participants With Proton Pump Inhibitor (PPI) and Other Gastric Protective Drug Utilization
Description: PPI and other gastric protective drug (defined as Histamine-2 receptor antagonists [H2RA], misoprostol, sucralfate, and others such as antacids) utilization.
Time Frame: Baseline through week 24 or ET
Population: ITT; any randomized participant who received at least one dose of study medication; N= number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3720 | 3718
Percentage of participants
  PPIs | 23.0 | 24.2
  H2RAs | 5.0 | 5.7
  Gastric protective agents | 0.9 | 1.0

15. Other Pre Specified Outcome: Percentage of Participants With Non-study Medication Utilization
Description: Non-study medication utilization associated with initial treatment defined as narcotic analgesics and acetaminophen use.
Time Frame: Baseline through week 24 or ET
Population: ITT; N= number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 3720 | 3718
Percentage of participants
  Acetaminophen | 6.8 | 6.5
  Acetylsalicylic acid (ASA) | 3.5 | 3.0
  NSAIDs | 12.8 | 13.3
  Opioids | 14.2 | 15.6

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib | nsNSAIDs
Serious Adverse Events (participants affected / at risk) | 99/3970 | 95/3951
Other Adverse Events (participants affected / at risk) | 962/3970 | 1163/3951
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=3970) | nsNSAIDs (N=3951)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Bezoar (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 10 | 7
Device dislocation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 1 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 3
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 3
Scrotal abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Vaginal abscess (Infections and infestations) | 0 | 1
Bone fragmentation (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood amylase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Musculoskeletal and connective tissue disorders) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 3
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Breast lump removal (Surgical and medical procedures) | 1 | 0
Colectomy (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Foot amputation (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 2
Spinal laminectomy (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=3970) | nsNSAIDs (N=3951)
Abdominal discomfort (Gastrointestinal disorders) | 30 | 52
Abdominal pain (Gastrointestinal disorders) | 37 | 59
Abdominal pain upper (Gastrointestinal disorders) | 37 | 60
Constipation (Gastrointestinal disorders) | 36 | 70
Diarrhoea (Gastrointestinal disorders) | 84 | 115
Dyspepsia (Gastrointestinal disorders) | 65 | 98
Gastritis (Gastrointestinal disorders) | 32 | 39
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 29 | 78
Nausea (Gastrointestinal disorders) | 65 | 112
Oedema peripheral (General disorders) | 50 | 67
Bronchitis (Infections and infestations) | 86 | 77
Sinusitis (Infections and infestations) | 75 | 88
Upper respiratory tract infection (Infections and infestations) | 112 | 75
Urinary tract infection (Infections and infestations) | 70 | 75
Fall (Injury, poisoning and procedural complications) | 44 | 64
Haemoglobin decreased (Investigations) | 59 | 84
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 | 73
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 43
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 29 | 39
Pain in extremity (Musculoskeletal and connective tissue disorders) | 59 | 47
Dizziness (Nervous system disorders) | 43 | 51
Headache (Nervous system disorders) | 67 | 83
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 41
Rash (Skin and subcutaneous tissue disorders) | 40 | 44
Hypertension (Vascular disorders) | 35 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.